CLINICAL TRIAL: NCT04518046
Title: A Phase 1/1b Study of Sitravatinib in Combination With Nivolumab and Ipilimumab in Patients With Advanced or Metastatic Clear-Cell Renal Cell Carcinoma or Other Solid Malignancies
Brief Title: Study of Sitravatinib, Nivolumab and Ipilimumab in Advanced or Metastatic Clear-Cell Renal Cell Carcinoma or Other Solid Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mirati Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 516-008
Record Dates: First submitted 2020-08-03; First posted 2020-08-19 (Actual); Last update posted 2024-06-05 (Actual); Status verified 2024-06

CONDITIONS: Clear-Cell Renal Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — sitravatinib; Nivolumab; Ipilimumab

STUDY DESIGN:
Intervention Model Description: Following the identification of the recommended dose of sitravatinib in combination with NIVO/IPI Phase 1 dose escalation, two Phase 1b dose expansion cohorts will enroll patients with ccRCC based on IMDC risk. All patients receive the same treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Phase 1: Dose Escalation (Experimental): Patients with poor- or intermediate-risk RCC with clear cell component for first-line treatment.
  Interventions: Drug: Sitravatinib; Drug: Nivolumab; Drug: Ipilimumab
- Phase 1b Dose Escalation Cohort A (Experimental): Patients with poor- or intermediate-risk RCC with clear cell component for first-line treatment
  Interventions: Drug: Sitravatinib; Drug: Nivolumab; Drug: Ipilimumab
- Phase 1b Dose Escalation Cohort B (Experimental): Patients with favorable-risk RCC with clear cell component for first-line treatment.
  Interventions: Drug: Sitravatinib; Drug: Nivolumab; Drug: Ipilimumab

INTERVENTIONS:
Drug: Sitravatinib — Sitravatinib is a small molecule inhibitor of receptor tyrosine kinases
  Other Names: MGCD516
Drug: Nivolumab — Nivolumab is a programmed death receptor-1 (PD-1) blocking antibody
  Other Names: OPDIVO
Drug: Ipilimumab — Ipilimumab is a CTLA-4 (cytotoxic T-lymphocyte-associated protein 4) blocking antibody
  Other Names: YERVOY

SUMMARY:
Study 516-008 is an open-label Phase 1 dose escalation/Phase 1b dose expansion study evaluating the safety and tolerability, clinical activity, and PK of sitravatinib in combination with nivolumab and ipilimumab for the treatment of ccRCC and potentially other solid tumor types.

DETAILED DESCRIPTION:
Sitravatinib is a spectrum-selective receptor tyrosine kinase (RTK) inhibitor that inhibits several closely related RTKs including the TAM family (Tyro3/Axl/MERTK), VEGFR2, KIT, and MET.

NIVO/IPI are monoclonal antibodies (mAbs) that inhibit the immune checkpoint proteins programmed death receptor-1 (PD-1) and cytotoxic T- lymphocyte antigen-4 (CTLA-4), respectively.

The current study is designed to evaluate the triple combination of sitravatinib plus NIVO/IPI in patients with solid tumor malignancies that have shown favorable responses to NIVO/IPI combinations in previous clinical trials. Combining sitravatinib and NIVO/IPI is predicted to have complementary effects in triggering a tumor-directed immune response.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of Clear-Cell Renal Cell Carcinoma (for initial cohorts under consideration)
* No prior treatment with systemic therapy (for initial cohorts under consideration)
* Adequate bone marrow and organ function

Exclusion Criteria:

* Known or suspected presence of other cancer
* Brain metastases (for initial cohorts under consideration)
* Carcinomatous meningitis
* Immunocompromising conditions
* Impaired heart function
* Active or prior documented autoimmune disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2020-08-11 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Frequency of patients experiencing treatment-emergent AEs | Through study completion, an average of 12 months
  Characterization of AEs by incidence, severity, timing, seriousness & relationship to study treatment

SECONDARY OUTCOMES:
Objective Response Rate (ORR) in accordance with RECIST v1.1 | Through duration of study, average of 10 months
  Frequency of patients experiencing an objective response
Duration of Response (DOR) | Through duration of study, average of 10 months
  Time in months from date of the first documentation of objective tumor response (CR or PR) to the first documentation of objective PD or to death due to any cause in the absence of documented PD
Progression-free Survival (PFS) | Through duration of study, average of 10 months
  Time from date of first study treatment to first PD or death due to any cause in the absence of documented PD

CONTACTS AND LOCATIONS:
Overall Officials: Curtis Chin, MD, Study Director — Mirati Therapeutics Inc.
Locations (1):
- MD Anderson, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Msaouel P, Yu K, Yuan Y, Chen J, Yan X, Karki M, Duan F, Sheth RA, Rao P, Sircar K, Shah AY, Zurita AJ, Genovese G, Li M, Yeh CC, Dang M, Han G, Chu Y, Hallin M, Olson P, Yang R, Slavin D, Der-Torossian H, Chin CD, Tannir NM, Wang L, Gao J. Sitravatinib in combination with nivolumab plus ipilimumab in patients with advanced clear cell renal cell carcinoma: a phase 1 trial. Nat Commun. 2025 Jan 10;16(1):578. doi: 10.1038/s41467-024-55642-8. PMID 39794332